CLINICAL TRIAL: NCT00214253
Title: Islet Transplantation in Type 1 Diabetic Patients Using a Steroid-free Immunosuppression Protocol and Thiazolidinedione Insulin Sensitizers
Brief Title: Islet Transplantation in Type 1 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001-529
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — 2,4-thiazolidinedione

ARMS (2):
- 1 (Experimental): Thiazolidinedione therapy
  Interventions: Drug: Thiazolidinedione
- 2 (No Intervention)

INTERVENTIONS:
Drug: Thiazolidinedione — Thiazolidinedione vs. no intervention with standard immunosuppression using Edmonton Protocol
  Arms: 1

SUMMARY:
Our hypothesis is that a successful clinical islet transplant program can be established at the University of Wisconsin using a steroid -free, sirolimus- and low dose tacrolimus - based immunosuppressive drug regimen (Edmonton protocol). We intend to answer the following research questions: 1) will treatment of islet transplant recipients with thiazolidinediones (i.e. pioglitazone) enhance post-transplant islet function and reduce the number of islets necessary to achieve adequate metabolic control? 2) which type 1 diabetic patients are optimal candidates for islet transplantation (i.e. islet transplant alone or islet after kidney transplantation)? 3) Can cadaver donor pancreases, which are ordinarily discarded and not used for pancreas transplantation be used for islet transplantation?

ELIGIBILITY:
Inclusion Criteria:

* 16 Type I insulin-dependent diabetic subjects ages 18-60,(8 who have received a prior kidney or liver transplant and have stable renal function, and 8 who have labile glucose regulation and who have failed a trial of intensive exogenous insulin therapy and who have preserved native renal function)

Exclusion Criteria:

* untreated proliferative diabetic retinopathy;
* HgbA1C >12%; creatinine clearance < 80 ml/minute or macroalbuminuria > 0.3 gm/24 hrs;
* presence of panel reactive antibodies >20%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
number of islets necessary to achieve adequate metabolic control | 5 years
post-transplant islet function | 5 years

SECONDARY OUTCOMES:
Suitability of cadaver donor pancreases for islet transplantation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jon Odorico, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States